CLINICAL TRIAL: NCT00327587
Title: An 8-week, Multicenter Study to Evaluate the Efficacy and Safety of the Combination of Valsartan/HCTZ/Amlodipine Compared to Valsartan/HCTZ, Valsartan/Amlodipine, and HCTZ/Amlodipine in Patients With Moderate to Severe Hypertension.
Brief Title: 8-week Study to Evaluate Safety and Efficacy of Various Combinations of Valsartan, HCTZ, and Amlodipine in Patients With Moderate to Severe Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVEA489A2302
Record Dates: First submitted 2006-05-16; First posted 2006-05-18 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Hypertension
Keywords: hypertension; valsartan; amlodipine; HCTZ
MeSH Terms: conditions — Hypertension | interventions — Amlodipine, Valsartan Drug Combination; Valsartan; Hydrochlorothiazide; Amlodipine

INTERVENTIONS:
Drug: Valsartan + amlodipine
Drug: Valsartan + HCTZ
Drug: Amlodipine + HCTZ
Drug: Valsartan + amlodipine + HCTZ

SUMMARY:
The purpose of this study is to determine the safety and efficacy of the various combinations of valsartan, HCTZ, and amlodipine in patients with moderate to severe hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate to severe hypertension (MSDBP ≥ 100 mmHg and < 120 mmHg, MSSBP ≥ 145 mmHg and < 200 mmHg).

Exclusion Criteria:

* Patients on two or more antihypertensive drugs with MSSBP ≥ 180 mmHg and/or MSDBP ≥ 110 mmHg at Visit 1.
* Patients on three or more antihypertensive drugs with MSDBP ≥ 90 mmHg and < 110 mmHg, and/or MSSBP ≥ 140 mmHg and < 180 mmHg at Visit 1.
* Patients on four or more antihypertensive drugs at Visit 1.
* Arm circumference > 42 cm for patients participating in ABPM.

Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2279 (Actual)
Dates: Start 2006-05; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline diastolic blood pressure after 8 weeks
Change from baseline systolic blood pressure after 8 weeks

SECONDARY OUTCOMES:
Blood pressure less than 140/90 mmHg after 8 weeks
Systolic blood pressure less than 140 mmHg or diastolic blood pressure less than 90 mmHg after 8 weeks
Diastolic blood pressure less than 90 mmHg or at least a 10 mmHg decrease after 8 weeks or systolic blood pressure less than 140 mmHg or at least a 15 mmHg decrease after 8 weeks
Ambulatory blood pressure and standing systolic and diastolic blood pressure measurements
Adverse events, serious adverse events, laboratory values, physical examinations, and vital signs for up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Principal Investigator — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals Corporation, East Hanover, New Jersey, United States

REFERENCES:
- [Derived] Calhoun DA, Lacourciere Y, Crikelair N, Jia Y, Glazer RD. Effects of demographics on the antihypertensive efficacy of triple therapy with amlodipine, valsartan, and hydrochlorothiazide for moderate to severe hypertension. Curr Med Res Opin. 2013 Aug;29(8):901-10. doi: 10.1185/03007995.2013.803057. Epub 2013 Jul 1. PMID 23721363
- [Derived] Lacourciere Y, Crikelair N, Glazer RD, Yen J, Calhoun DA. 24-Hour ambulatory blood pressure control with triple-therapy amlodipine, valsartan and hydrochlorothiazide in patients with moderate to severe hypertension. J Hum Hypertens. 2011 Oct;25(10):615-22. doi: 10.1038/jhh.2010.115. Epub 2011 Jan 20. PMID 21248785